CLINICAL TRIAL: NCT00448396
Title: An Open Label Phase I Study to Evaluate the Effects of Patupilone on the Pharmacokinetics and Pharmacodynamics of Warfarin in Patients With Advanced Malignancies
Brief Title: Evaluate the Effects of Patupilone on the Pharmacokinetics and Pharmacodynamics of Warfarin in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2120
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Malignancies
Keywords: Cancer; EPO; Patupilone; Solid tumors; Advanced malignancies
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

ARMS (1):
- Patupilone (Experimental)
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
To evaluate the effects of patupilone on the pharmacokinetics of warfarin in patients with advanced malignancies.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years of age
* Life expectancy ≥3 months
* Histologically documented advanced solid tumors which have progressed after standard systemic therapy or for which standard systemic therapy does not exist
* Agents containing warfarin or heparin must be discontinued 7 days prior to enrollment in the study

Exclusion criteria

* History of/or active bleeding disorders
* Known hypersensitivity to warfarin or related compounds
* The use of vitamin K
* Central lines that require anticoagulant maintenance
* The use of agents containing warfarin and heparin
* Known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of patupilone on the pharmacokinetics of warfarin in patients with advanced malignancies.

SECONDARY OUTCOMES:
To evaluate the effects of patupilone on the pharmacodynamics of warfarin in patients with advanced malignancies.
Safety and tolerability of patupilone when administered concomitantly with warfarin in patients with advanced malignancies will be assessed by AE's, SAE's and safety labs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- San Antonio, Texas, United States